CLINICAL TRIAL: NCT03388619
Title: A Phase I Trial of Highly Conformal, Hypofractionated, Focally Dose Escalated Post-Prostatectomy Radiotherapy
Brief Title: Highly Conformal, Hypofractionated, Focally Dose Escalated Post-Prostatectomy Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180028; 18-C-0028
Record Dates: First submitted 2017-12-30; First posted 2018-01-03 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cancer Of Prostate; Prostate Neoplasms; Prostate Cancer; Neoplasms of Prostate; Prostatic Cancer
Keywords: Rising PSA; No evidence of metastatic disease; Entire Prostate Bed; Quality of Life; Irradiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tomography, X-Ray Computed; Multiparametric Magnetic Resonance Imaging; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm 1/Prostate Bed with Integrated Boost (Experimental): Prostate bed with integrated boost.
  Interventions: Radiation: Prostate bed with integrated boost; Diagnostic Test: Whole Body Bone Scan; Diagnostic Test: 18F-NaF PET Imaging; Diagnostic Test: CT; Diagnostic Test: mpMRI; Drug: ADT
- Arm 2/Prostate Bed Irradiation Only (Experimental): Prostate bed irradiation only.
  Interventions: Radiation: Prostate bed irradiation only; Diagnostic Test: Whole Body Bone Scan; Diagnostic Test: 18F-NaF PET Imaging; Diagnostic Test: CT; Diagnostic Test: mpMRI; Drug: ADT

INTERVENTIONS:
Radiation: Prostate bed with integrated boost — Radiation will be delivered at an escalated dose to areas of recurrent prostate cancer identified on imaging and a reduced dose will be delivered to the entire prostate bed.
  Arms: Arm 1/Prostate Bed with Integrated Boost
Radiation: Prostate bed irradiation only — Radiation will be delivered to the prostate bed only.
  Arms: Arm 2/Prostate Bed Irradiation Only
Diagnostic Test: Whole Body Bone Scan — At screening, if required by clinician.
Diagnostic Test: 18F-NaF PET Imaging — At screening, if required by clinician.
  Other Names: Fluorine 18-sodium fluoride positron emission tomography
Diagnostic Test: CT — Computed tomography of the abdomen and pelvis if clinically indicated at screening, with oral and intravenous contrast.
  Other Names: Computed tomography
Diagnostic Test: mpMRI — mpMRI of the prostate bed at screening and 6 month follow up.
  Other Names: Multiparametric magnetic resonance imaging
Drug: ADT — After enrollment if clinically indicated (i.e., anti-androgen, gonadotropin releasing hormone agonist, or combination of both).
  Other Names: androgen deprivation therapy

SUMMARY:
Background:

Sometimes prostate cancer comes back after a person's prostate is removed. In this case, radiation is a common treatment. Radiation kills prostate cancer cells. It can be very effective. It is usually given in short doses almost every day for 6 or 7 weeks. Researchers want to see if a shorter schedule can be as effective. They want to see if that causes the same or fewer side effects. Usually, radiation is used to treat the entire area where the prostate was before surgery. In some patients, an area of tumor can be seen on scans. Researchers are also trying to see if they can give less dose to the area usually treated with radiation if the full dose is given to the tumor seen on scans.

Objective:

To find the shortest radiation schedule that people can tolerate without strong side effects.

Eligibility:

People at least 18 years old who have had a prostatectomy and will get radiation.

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests
* Scan that uses a small amount of radiation to make a picture of the body
* Scan that uses a magnetic field to make an image of the body
* Participants will provide documents that confirm their diagnosis.
* Participants may have a scan of the abdomen and pelvis.

Before they start treatment, participants will have another physical exam and blood tests.

Participants will get radiation each day Monday through Friday. Treatment may last 2, 3, or 4 weeks.

Participants may provide a tissue sample from a previous procedure for research.

Participants will answer questions about their general well-being and function.

About 4-5 weeks after they finish radiation treatment, participants will have a follow-up visit. They will be examined and give a blood sample. They will have 6 follow-up visits for the next 2 years.

DETAILED DESCRIPTION:
BACKGROUND:

Prostate cancer that recurs after prostatectomy (rising prostate-specific antigen (PSA) with no evidence of metastatic disease is often treated with radiation to the entire prostate bed to a dose of 66-72 Gray (Gy) over 6-7 weeks. This treatment can provide PSA control in approximately 75% of patients but may have associated genitourinary and gastrointestinal toxicity due to irradiation of the rectum, small bowel, and bladder. Imaging of prostate cancer has improved to the extent that recurrent disease is often identified in the prostate bed or in other pelvic sites. The current standard is to irradiate the entire prostate bed to the total dose. This trial will test the tolerability of accelerated treatment designed to yield a similar rate of late toxicity. In addition, in patients with visible tumor, it will test the feasibility of delivering a lower dose to the prostate bed and an integrated boost (simultaneous) to the visible tumor to allow a higher dose to visible tumor than can be delivered with standard approaches.

OBJECTIVE:

- Define the maximum tolerated dose (MTD) hypofractionation of image guided, focally dose escalated post-prostatectomy radiation.

ELIGIBILITY:

* PSA recurrence after prostatectomy or indications for adjuvant radiation after prostatectomy.
* No evidence of distant metastases of prostate cancer (pelvic lymph nodes are allowed).
* Age greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1

DESIGN:

This is a Phase I trial of hypofractionated focal dose escalation with reduced dose prostate bed irradiation using image and pathologic guidance. The prostate bed will be treated with hypofractionated radiation and areas in the prostate bed or pelvis shown to have tumor on biopsy or with advanced imaging studies will be treated with an integrated boost to visible tumor. The treatment duration will be decreased sequentially in three Dose Level groups. Quality of life and functional outcomes such as urine, bowel, and erectile function will be assessed with questionnaires. A maximum of 48 patients will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed adenocarcinoma of the prostate.
* Indications for post-prostatectomy radiation exist:

  * Disease progression (detectable prostate-specific antigen (PSA) on two measurements obtained at least one month apart) or
  * indications for adjuvant radiation exist (if undetectable PSA): pathologic T3, T4, N+ disease or positive margins (within 1 year of prostatectomy).
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 60)
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Radiation is teratogenic; thus, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and up to 120 days after the last radiation. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Human immunodeficiency virus (HIV) positive patients are included if CD4+ (cytotoxic T cells) T-cell count > 200 cells/uL; on stable antiretroviral therapy for > 1 year with HIV viral load <200 copies/mL, and no history of opportunistic infections in > 1 year.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents concurrently.
* Documented metastases of prostate cancer outside of the pelvis (pelvic lymph nodes are allowed only if within the prostate bed region).
* History of radiation that would overlap with the intended treatment to the prostate bed.
* Known contraindications to radiation such as inflammatory bowel disease, active systemic lupus or scleroderma, or radiation hypersensitivity syndrome (Ataxia Telangiectasia or Fanconi's Anemia)
* Subjects with any coexisting medical or psychiatric condition which, in the opinion of the Investigator likely to interfere with study procedures and/or results.
* Medically indicated use of known radiosensitizing drugs (such as protease inhibitors)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2025-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Shaikh T, Li T, Handorf EA, Johnson ME, Wang LS, Hallman MA, Greenberg RE, Price RA Jr, Uzzo RG, Ma C, Chen D, Geynisman DM, Pollack A, Horwitz EM. Long-Term Patient-Reported Outcomes From a Phase 3 Randomized Prospective Trial of Conventional Versus Hypofractionated Radiation Therapy for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):722-731. doi: 10.1016/j.ijrobp.2016.12.034. Epub 2016 Dec 28. PMID 28244407
- [Background] Christie DR, Sharpley CF, Bitsika V. Why do patients regret their prostate cancer treatment? A systematic review of regret after treatment for localized prostate cancer. Psychooncology. 2015 Sep;24(9):1002-11. doi: 10.1002/pon.3776. Epub 2015 Mar 1. PMID 25728586
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0028.html

RESULTS

PARTICIPANT FLOW:
Groups:
- LEVEL 1/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions: LEVEL 1/ COHORT 1: Recurrent tumor visible; prostate bed with integrated boost. 20 fractions: Dose to prostate bed 45.8 Gray (Gy) in 2.29 Gy fractions; Dose to tumor 60.4 Gy in 3.02 Gy fractions.
- LEVEL 2/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions: LEVEL 2/ COHORT 1: Recurrent tumor visible, prostate bed with integrated boost. 15 fractions: Dose to prostate bed 41.85 Gray (Gy) in 2.79 Gy fractions; Dose to tumor 54.6 Gy in 3.64 Gy fractions.
- LEVEL 3/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions: LEVEL 3/ COHORT 1: Recurrent tumor visible, prostate bed with integrated boost. 10 fractions: Dose to prostate bed 36.4 Gray (Gy) in 3.64 Gy fractions; Dose to tumor 47.1 Gy in 4.71 Gy fractions.
- LEVEL 1/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions: LEVEL 1/ COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 20 fractions: Dose to prostate bed 56.4 Gray (Gy) in 2.82 Gy fractions.
- LEVEL 2/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions: LEVEL 2/ COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 15 fractions: Dose to prostate bed 51.2 Gray (Gy) in 3.41 Gy fractions.
- LEVEL 3/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions: LEVEL 3/ COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 10 fractions: Dose to prostate bed 44.2 Gray (Gy) in 4.42 Gy fractions.
Period: Overall Study
Arm/Group | LEVEL 1/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions
Started | 3 | 3 | 9 | 3 | 3 | 9
Follow-up period completed. | 3 | 3 | 5 | 3 | 3 | 8
Completed | 3 | 3 | 9 | 3 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEVEL 1/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/ COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/ COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions | Total
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 3 | 9 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 1 | 0 | 4 | 10
  >=65 years | 2 | 2 | 6 | 2 | 3 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.63 (7.35) | 67.4 (3.02) | 67.04 (7.51) | 67.63 (9.87) | 70.87 (1.61) | 64.32 (10.4) | 66.56 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 9 | 3 | 3 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 9 | 3 | 3 | 8 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 0 | 1 | 2 | 8
  White | 1 | 3 | 6 | 3 | 2 | 7 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 9 | 3 | 3 | 9 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Radiation Dose to Prostate Bed and Dose to Tumor Reported in Gray (Gy)
Description: Maximum tolerated dose (MTD) of image guided hypofractionated, focally dose escalated post-prostatectomy radiation is defined as the dose level at which no more than 1 of up to 6 participants experience dose limiting toxicity (DLT) during the DLT period, and the dose below that at which at least 2 (of ≤6) participants have DLT as a result of treatment. A DLT is defined as any of the following: Grade 3 rectal, small bowel, or urinary toxicity that does not resolve to Grade 2 or less within 4 days with appropriate medical management. Other grade 3 in-field toxicities attributable to radiation that does not resolve to Grade 2 or less within 4 days with appropriate medical management. And delays of more than one week in completing radiation treatment due to toxicity.
Time Frame: 3 weeks after radiation
Population: 12/30 expansion group participants (6 in Recurrent Tumor Visible: Level 3 Cohort 1, and Recurrent Tumor NOT Visible: Level 3 Cohort 2) were not assessed for MTD and included in the analysis.
Measure: Number; unit: Gray (Gy)
Groups:
- All Participants With Recurrent Tumor Visible: All participants with recurrent tumor visible assessed for MTD.
  Level 1 Cohort 1, Level 2 Cohort 1, and Level 3 Cohort 1:
  Recurrent tumor visible, prostate bed with integrated boost. 10 fractions: Dose to prostate bed 36.4 Gray (Gy) in 3.64 Gy fractions; Dose to tumor 47.1 Gy in 4.71 Gy fractions.
- All Participants With Recurrent Tumor NOT Visible: All participants with recurrent tumor NOT visible assessed for MTD.
  Level 1 Cohort 2, Level 2 Cohort 2, and Level 3 Cohort 2:
  Recurrent tumor NOT visible, prostate bed irradiation only. 10 fractions: Dose to prostate bed 44.2 Gray (Gy) in 4.42 Gy fractions.
Arm/Group | All Participants With Recurrent Tumor Visible | All Participants With Recurrent Tumor NOT Visible
Number analyzed (Participants) | 9 | 9
Gray (Gy)
  Dose to prostate bed | 36.4 | 44.2
  Dose to tumor: number analyzed (Participants) | 9 | 0
  Dose to tumor | 47.1 |

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Radiation Dose to Prostate Bed and Dose to Tumor Reported in Fractions
Description: as for outcome 1
Time Frame: 3 weeks after radiation
Population: as for outcome 1
Measure: Number; unit: Fractions
Arm/Group | All Participants With Recurrent Tumor Visible | All Participants With Recurrent Tumor NOT Visible
Number analyzed (Participants) | 9 | 9
Fractions
  Dose to prostate bed | 3.64 | 4.42
  Dose to tumor: number analyzed (Participants) | 9 | 0
  Dose to tumor | 4.71 |

3. Secondary Outcome: Biochemical Progression Free Survival (bPFS)
Description: bPFS is defined as the duration of time from start of treatment to time of prostate-specific antigen (PSA) progression or death, whichever occurs first. PSA progression (also known as biochemical failure) is defined based on elevation of PSA beyond 0.1 ng/dL. Kaplan-Meier survival analysis and effects of clinical variables on bPFS will be assessed by the Cox proportional hazards model.
Time Frame: 1 and 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Proportion of Participants That Have Improvement in Quality of Life After Treatment
Description: The quality-of-life scores will be summarized at baseline and for each visit. Linear mixed effects model will be used to model quality of life scores at baseline and during and after treatment in which random intercept and random slope are used to account for participant-specific trajectory of quality-of-life scores.
Time Frame: 1 and 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Sexual Health Inventory for Men (SHIM)
Description: Participants completed a 6-question questionnaire to assess erectile dysfunction.
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: American Urologic Association Symptom Index Score (AUA-SI)
Description: The AUA-SI is used to measure radiation morbidity and to make treatment decisions.
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression Short Form (SF) 4a:
Description: Participants complete a form to assess negative mood (i.e., sadness, guilt), views of self (i.e., self-criticism, worthlessness) social cognition (loneliness, interpersonal alienation), decreased positive effect, and decreased engagement (loss of interest, meaning, and purpose) and are scored using item-level calibrations.
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety Short Form (SF) 4a:
Description: Participants complete a form and rate anxiety such as fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness).
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) - Psychosocial Impact Positive Short Form (SF) 4a
Description: Participants complete a form to assess positive psychosocial (emotional and social) outcomes of illness.
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Decision Regret Scale (DRS)
Description: The DRS is a 5-item scale measuring distress or remorse after a health case decision. The score correlated with satisfaction with the decision (r=-0.40 to -0.60), decisional conflict (r=0.31 to 0.52), and overall rated quality of life (r=-0.25 to -0.27).
Time Frame: 2 years after treatment
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Grade 2-5 Serious and/or Non-serious Adverse Events Unlikely, Probably, Possibly and Definitely Attributable to Research
Description: Grade 2-5 serious and/or non-serious adverse events attributable to protocol treatment. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 2 is moderate. Grade 3 is serious. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: 3 weeks after radiation
Measure: Number; unit: adverse events
Groups:
- LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions: LEVEL 1/COHORT 1: Recurrent tumor visible; prostate bed with integrated boost. 20 fractions: Dose to prostate bed 45.8 Gray (Gy) in 2.29 Gy fractions; Dose to tumor 60.4 Gy in 3.02 Gy fractions.
- LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions: LEVEL 2/COHORT 1: Recurrent tumor visible, prostate bed with integrated boost. 15 fractions: Dose to prostate bed 41.85 Gray (Gy) in 2.79 Gy fractions; Dose to tumor 54.6 Gy in 3.64 Gy fractions.
- LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions: LEVEL 3/COHORT 1: Recurrent tumor visible, prostate bed with integrated boost. 10 fractions: Dose to prostate bed 36.4 Gray (Gy) in 3.64 Gy fractions; Dose to tumor 47.1 Gy in 4.71 Gy fractions.
- LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions: LEVEL 1/COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 20 fractions: Dose to prostate bed 56.4 Gray (Gy) in 2.82 Gy fractions.
- LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions: LEVEL 2/COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 15 fractions: Dose to prostate bed 51.2 Gray (Gy) in 3.41 Gy fractions.
- LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions: LEVEL 3/COHORT 2: Recurrent tumor NOT visible, prostate bed irradiation only. 10 fractions: Dose to prostate bed 44.2 Gray (Gy) in 4.42 Gy fractions.
Arm/Group | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 3 | 9
adverse events
  Grade 2-5 Serious | 0 | 0 | 0 | 0 | 0 | 0
  Grade 2 Unlikely Related - Skin and subcutaneous tissue disorders - Other, specify | 1 | 0 | 0 | 0 | 0 | 0
  Grade 2 Unlikely Related Hemorrhoids | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Unlikely Related Testicular pain | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Unlikely Related Testicular disorder | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Possibly Related Urinary tract obstruction | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 Possibly Related Flatulence | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Possibly Related Hemorrhoids | 0 | 0 | 0 | 0 | 0 | 2
  Grade 2 Possibly Related Diarrhea | 0 | 0 | 0 | 1 | 0 | 1
  Grade 2 Possibly Related Skin infection | 0 | 0 | 0 | 0 | 0 | 1
  Grade 2 Probably Related Rectal hemorrhage | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Probably Related - Urinary urgency | 1 | 0 | 0 | 0 | 0 | 1
  Grade 2 Probably Related Proctitis | 0 | 2 | 3 | 0 | 2 | 6
  Grade 2 Probably Related Urinary urgency | 0 | 1 | 0 | 0 | 1 | 0
  Grade 2 Probably Related Diarrhea | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Probably Related Flatulence | 0 | 0 | 2 | 0 | 0 | 0
  Grade 2 Probably Related Hemorrhoids | 0 | 1 | 1 | 0 | 0 | 5
  Grade 2 Probably Related Cystitis noninfective | 0 | 0 | 0 | 0 | 1 | 1
  Grade 2 Probably Related Urinary frequency | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Probably Related Urinary incontinence | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Probably Related Proctitis | 0 | 0 | 1 | 0 | 0 | 0
  Grade 3 Probably Related Urinary incontinence | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Probably Related Cystitis noninfective | 0 | 0 | 0 | 0 | 1 | 0
  Grade 2 Definitely Related Flatulence | 0 | 0 | 1 | 0 | 0 | 0
  Grade 2 Definitely Related Proctitis | 0 | 0 | 3 | 0 | 0 | 4

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 3 | 9
Participants | 3 | 3 | 8 | 3 | 3 | 9

13. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: A DLT is defined as any of the following: Grade 3 rectal, small bowel, or urinary toxicity that does not resolve to Grade 2 or less within 4 days with appropriate medical management. Other grade 3 in-field toxicities attributable to radiation that does not resolve to Grade 2 or less within 4 days with appropriate medical management. And delays of more than one week in completing radiation treatment due to toxicity.
Time Frame: 3 weeks after radiation
Measure: Count of Participants; unit: Participants
Arm/Group | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions
Number analyzed (Participants) | 3 | 3 | 9 | 3 | 3 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 25 months.
Arm/Group | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 0/3 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/9 | 1/3 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 8/9 | 3/3 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions (N=3) | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions (N=3) | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions (N=9) | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions (N=3) | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions (N=3) | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions (N=9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEVEL 1/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 20 Fractions (N=3) | LEVEL 2/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 15 Fractions (N=3) | LEVEL 3/COHORT 1: Recurrent Tumor Visible; Prostate Bed With Integrated Boost - 10 Fractions (N=9) | LEVEL 1/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 20 Fractions (N=3) | LEVEL 2/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 15 Fractions (N=3) | LEVEL 3/COHORT 2: Recurrent Tumor NOT Visible; Prostate Bed Irradiation Only - 10 Fractions (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, palpitations, PVC?s, dizziness, history of chest pain (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis noninfective (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (5)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (7) | 0 (0) | 1 (1) | 3 (4)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, fecal urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, passing stool with gas (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (9)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, Right great toe "Turf toe" (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, Right left second toe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Proctitis (Gastrointestinal disorders) | 0 (0) | 2 (4) | 6 (7) | 0 (0) | 2 (3) | 9 (17)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, Post Traumatic Stress Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, weak stream (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, Climacturia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, Internal pulling sensation suprapubic (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Gluteal cleft fissure (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hyperpigmented macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Tinea cruris (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, contact dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 3 (4)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03388619/Prot_SAP_002.pdf
  • Informed Consent Form (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03388619/ICF_001.pdf